CLINICAL TRIAL: NCT05754879
Title: Congenital Cytomegalovirus Infection by Detection of the Virus in the Saliva of Newborns at Particular Risk: A Retrospective Population-based Study Between February 2019 and December 2021 at the Regional Maternity Hospital of Nancy
Brief Title: Diagnosis of Congenital Cytomegalovirus Infection in Newborn With Particular Risk
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: 2022PI027
Record Dates: First submitted 2023-02-13; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Congenital Cytomegalovirus Infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital CMV infection is the leading cause of non-genetic deafness and neurodevelopmental disorders. Its prevalence in France is estimated between 0.3% and 1% of births depending on the study.

Congenital infection is symptomatic in 10% of cases with a large clinical spectrum with different degree of severity. These sequelae develop progressively and fluctuate, which justifies prolonged follow-up of children for several years, even if they are asymptomatic at birth.

There is yet no treatment with AMM in neonates or pregnant women. In France, screening for congenital CMV infection is widely debated. It remains oriented to certain newborns considered at risk or depending on their symptoms and varies with the practices of each Neonatology or Maternity Hospital.

In the Regional Maternity of Nancy, a new screening protocol for congenital CMV infection was implemented from early 2019.

It is based on screening by non-invasive salivary test (CMV PCR) in newborns at particular risk who are included in a registry open for this screening.

The aim of this research was to assess the relevance of the proposed criteria in the Protocol for defining a population at risk of congenital CMV infection thus qualifying for CMV screening. The secondary endpoints are the modalities of the screening test, the evaluation of each risk factor for infection, and the study of affected patients (symptoms, therapeutic intervention, neurological and auditory outcome).

ELIGIBILITY:
Inclusion Criteria:

* Newborn born between Bebruary 2019 and December 2021 in the Regional Maternity Hospital of Nancy
* Patients who were screened for congenital CMV infection by salivary PCR

Exclusion Criteria:

* No one

Max Age: 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All NewBorn born between January 2019 and December 2021 who have had Screening Congenital Cytomegalovirus Infection by PCR in saliva
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Relevance of the Protocol for defining a population at risk | baseline
  Comparison between Prevalence in the targeted population and Prevalence in the general Population

SECONDARY OUTCOMES:
Modalities of realisation of screening test | baseline
  Test by PCR in saliva and appropriate indications
Maternal CMV infection as a Risk Factor for Congenital CMV Infection | baseline
  Association between Maternal infection and Neonatal CMV infection
Hypotrophy as a Risk Factor for Congenital CMV Infection | baseline
  Association of a Neonatal weight below the 10th centile and Neonatal CMV infection
Microcephaly as a Risk Factor for Congenital CMV Infection | baseline
  Association of a Neonatal head circumference below the 10th centile and Neonatal CMV infection
Any foetal ultrasound abnormality as a Risk Factor for Congenital CMV Infection | baseline
  Association of any abnormality at fetal ultrasound examination and Neonatal CMV infection
Presence of Hepatomegaly or splenomegaly as a Risk Factor for Congenital CMV Infection | baseline
  Association of hepatomegaly or splenomegaly and Neonatal CMV infection
Any neurological abnormality as a Risk Factor for Congenital CMV Infection | baseline
  Any neurological abnormality at clinical examination as a Risk Factor for Congenital CMV Infection
Any blood count cell abnormality as a Risk Factor for Congenital CMV Infection | baseline
  Any blood count cell abnormality at biological check up as a Risk Factor for Congenital CMV Infection
Biological hepatic abnormality as a Risk Factor for Congenital CMV Infection | baseline
  Any biological hepatic abnormality at biological check up as a Risk Factor for Congenital
Hearing abnormality as a Risk Factor for Congenital CMV Infection | baseline
  Failure at hearing screening as a Risk Factor for Congenital CMV Infection
Hypotrophy as a consequence of diagnosed Congenital CMV Infection | baseline
  Association of a birth weight below the 10th centile with a diagnosed Neonatal CMV infection
Microcephaly as a consequence of diagnosed Congenital CMV Infection | baseline
  Association of a Neonatal head circumference below the 10th centile with a diagnosed Neonatal CMV infection
Presence of Hepatomegaly or splenomegaly as a Risk Factor for Congenital CMV Infection | Baseline
  Association of an hepatomegaly or spenomegly with a diagnosed Neonatal CMV infection
Any neurological abnormality as a consequence of Congenital CMV Infection | baseline
  Association of a neurological abnormality at clinical examniation with a diagnosed Neonatal CMV infection
Any blood count cell abnormality as a consequence of Congenital CMV Infection | baseline
  Association of any blood count cell abnormality with a diagnosed Neonatal CMV infection
Biological hepatic abnormality as a consequence of Congenital CMV Infection | baseline
  Association of any biological hepatic abnormality with a diagnosed Neonatal CMV infection
Hearing abnormality as a consequence of Congenital CMV Infection | baseline
  Association of failure at hearing screening with a diagnosed Neonatal CMV infection

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Hospital CHRU, Nancy, France